CLINICAL TRIAL: NCT01259752
Title: Prospective Randomized Study of Compression Stockings in Ankle Sprain in Adults
Brief Title: Compression Stockings in Ankle Sprain
Acronym: CASED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pierre and Marie Curie University (Other); Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P080603
Record Dates: First submitted 2010-09-23; First posted 2010-12-14 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2010-06

CONDITIONS: Ankle Sprain
Keywords: Trauma; ankle sprain; emergency; compression stocking
MeSH Terms: conditions — Ankle Injuries; Wounds and Injuries; Emergencies | interventions — Stockings, Compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- compression stockings (Experimental)
  Interventions: Device: compression stockings
- standard non compressive stockings (Placebo Comparator)
  Interventions: Other: standard non compressive stockings

INTERVENTIONS:
Device: compression stockings — compression stockings
  Arms: compression stockings
Other: standard non compressive stockings — standard non compressive stockings
  Arms: standard non compressive stockings

SUMMARY:
This is a multicenter prospective randomized superiority controlled trial comparing leg stockings and standard care to standard care of ankle sprain and testing the hypothesis that compression stockings enable to reduce the median of recovery from ankle sprain by at least 6 days.

DETAILED DESCRIPTION:
Introduction: Ankle sprain is a frequently encountered trauma lesion in emergency departments and is associated with important health expenses. However, appropriate care of this trauma lesion remains a matter of debate.

Hypothesis: The tested hypothesis is that compression stockings enable to reduce the median of recovery from ankle sprain by at least 6 days.

Main end point: Delay to recovery of normal painless walking, without any analgesic drug consumption.

Secondary end points : Pain at rest and during walking using a visual analog pain scale, bimalleolar and middle-feet perimeters, number of days with analgesic drug consumption, observance analysis, patient's tolerance using a visual analog scale, delay to recover sport activities in the subgroup of patients having a regular sport activity.

Methods: Multicenter Prospective randomized superiority controlled trial comparing leg stockings and standard care to standard care of ankle sprain. Standard care include the RICE (Rest, Ice, Compression, Elevation) protocol at admission, immobilization with ankle bracing (3 to 6 week duration according to severity and clinical course), recommendation for walking (no weight baring, partial weight bearing, total weight bearing), administration of analgesic drugs. The medical device tested in the present study is class II compressive stockings (compression between 15 and 20 mmHg).

Number of patients: With an alpha risk of 5%, a beta risk of 5%, 70 patients should be included in each group to be able to detect a 6 day difference in the delay of recovery, defined as normal painless walking without any analgesic drug consumption, taking into consideration 10% of patients lost during follow up.

Criteria for inclusion: Recent (<48h) ankle sprain without fracture and without other traumatic lesions in adult patients aged between 18 and 55 years. Patients with limb arterial disease, diabetes, or any diseases expected to potentially interfere with recovery of walking, are excluded as well as pregnant women.

Study schedule: Inclusion during first visit to the emergency department, then at day 7, 15-21, 30-45, and 90. Phone call interviews are performed to define the more appropriate timing of the visits.

ELIGIBILITY:
Inclusion Criteria:

* Recent (<48h) ankle sprain without fracture and without other traumatic lesions in adult patients aged between 18 and 55 years.

Exclusion Criteria:

* Patients with limb arterial disease, diabetes, or any diseases expected to potentially interfere with recovery of walking, are excluded as well as pregnant women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Delay to recovery of normal painless walking, without any analgesic drug consumption. | up to 90 days

SECONDARY OUTCOMES:
Pain at rest using a visual analog pain scale | at each follow-up visit (D-7, D-15 to 21, D-30 to 45)
Bimalleolar perimeter | at each follow-up visit (D-7, D-15 to 21, D-30 to 45)
Number of days with analgesic drug consumption | at each follow-up visit (D-7, D-15 to 21, D-30 to 45)
Observance analysis | at each follow-up visit (D-7, D-15 to 21, D-30 to 45)
  Number of days actually wearing compression stocking and ankle bracing and taking analgesic drugs
Delay to recover sport activities in the subgroup of patients having a regular sport activity | at each follow-up visit (D-7, D-15 to 21, D-30 to 45) and at the last follow-up visit (D-90)
Pain during walking using a visual analog pain scale | at each follow-up visit (D-7, D-15 to 21, D-30 to 45)
middle-feet perimeter | at each follow-up visit (D-7, D-15 to 21, D-30 to 45)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Hausfater, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Pitié Salpetriere hospital, Paris, France

REFERENCES:
- [Derived] Bendahou M, Khiami F, Saidi K, Blanchard C, Scepi M, Riou B, Besch S, Hausfater P. Compression stockings in ankle sprain: a multicenter randomized study. Am J Emerg Med. 2014 Sep;32(9):1005-10. doi: 10.1016/j.ajem.2014.05.054. Epub 2014 Jun 12. PMID 25043629